CLINICAL TRIAL: NCT05105737
Title: Retrospective Analysis of Degenerative Scoliosis Corrections by Posterior Instrumentation
Brief Title: Degenerative Scoliosis
Acronym: DS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7962
Record Dates: First submitted 2021-10-20; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Degenerative Scoliosis
Keywords: Degenerative Scoliosis; Degenerative lumbar scoliosis; Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Several deformities of the spine exist such as degenerative lumbar scoliosis. These deformities can generate functional discomfort and limit the patient's quality of life.

In the event of severe trunk imbalance and progression of the deformity, operative correction of the spinal deformity by instrumentation and posterior arthrodesis may be indicated.

Surgical techniques and instrumentation have evolved over the past 5 years. These changes in surgical strategies have a potential impact on the patient's quality of life and the correction results in the medium and long term.

The aim of the study is the analysis of surgical corrections obtained and radiological changes over time with classic 2-rod techniques versus modern 4-rod instrumentation techniques

ELIGIBILITY:
Inclusion criteria:

* Major subjects> 18 years old
* Subject with a surgical indication for arthrodesis and surgical correction of degenerative scoliosis
* Subject not having expressed his opposition, after information, to the reuse of his data for the purposes of this research.

Exclusion criteria:

* Subject having expressed opposition to participating in the study
* Subject under guardianship or guardianship
* Subject under safeguard of justice

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subject with a surgical indication for arthrodesis and surgical correction of degenerative scoliosis
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-10-29 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03-29 (Estimated)

PRIMARY OUTCOMES:
Retrospective analysis of degenerative scoliosis corrections by posterior instrumentation | Files analysed retrospectively from January 01, 2010 to December 31, 2010 will be examined]

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Chirurgie du Rachis - Hôpitaux Universitaires de Strasbourg, Strasbourg, France